CLINICAL TRIAL: NCT00560599
Title: A 2X2 Phase III Open-label Clinical Trial of Therapy for Patients With Recurrent Methicillin Resistant Staphylococcus Aureus Infections: Topical Nasal & Body Decolonization and/or Environmental Decontamination vs. Standard of Care
Brief Title: A Randomized Clinical Trial to Prevent Recurrent CA-MRSA Infection
Acronym: PRIMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: loren g miller (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor-Investigator, loren g miller, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 12550-01; KPSC IRB: 4714; CDC: 1U01CI000384-01
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Methicillin Resistant Staphylococcus Aureus Skin Infections
Keywords: MRSA; Methicillin Resistant Staphylococcus aureus; Staphylococcus aureus; Skin Infections; Body Decolonization; Environmental Decolonization
MeSH Terms: conditions — Staphylococcal Infections; Cellulitis | interventions — Mupirocin; Chlorhexidine; Disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Standard of care (No Intervention): Standard of care (no body decolonization regimen) and Standard of care (no environmental decolonization regimen)
- 2: Body decolonization regimen (Experimental): Body decolonization regimen and Standard of care (no environmental decolonization regimen)
  Interventions: Drug: mupirocin and chlorhexidine
- 3 Environmental decolonization regimen (Experimental): Standard of care (no body decolonization regimen) and Environmental decolonization regimen
  Interventions: Behavioral: household cleaning and disinfection
- 4 Body and Environmental decolonization regimens (Experimental): Body decolonization regimen and Environmental decolonization regimen
  Interventions: Drug: mupirocin, chlorhexidine, & household cleaning/disinfection

INTERVENTIONS:
Drug: mupirocin and chlorhexidine — Mupirocin (Bactroban Nasal): twice a day for 7 days, apply one pea-sized amount of Bactroban Nasal ointment directly into one nostril and another pea-sized amount for the other nostril.
  Chlorhexidine (Hibiclens): once a day for 14 days, rinse body with chlorhexidine.
  Arms: 2: Body decolonization regimen
Behavioral: household cleaning and disinfection — Environmental cleaning with topical ethanol and laundering of clothes and linen.
  Arms: 3 Environmental decolonization regimen
Drug: mupirocin, chlorhexidine, & household cleaning/disinfection — Mupirocin (Bactroban Nasal): twice a day for 7 days, apply one pea-sized amount of Bactroban Nasal ointment directly into one nostril and another pea-sized amount for the other nostril.
  Chlorhexidine (Hibiclens): once a day for 14 days, rinse body with chlorhexidine.
  Environmental cleaning with topical ethanol and laundering of clothes and linen.
  Arms: 4 Body and Environmental decolonization regimens

SUMMARY:
This clinical trial tests the hypotheses that 1) body decolonization of patients with recurrent community-associated (CA) MRSA infections and their household members and 2) environmental decolonization of the patients' households will significantly reduce the likelihood of recurrent CA-MRSA infection.

DETAILED DESCRIPTION:
Staphylococcus aureus is a ubiquitous pathogen, and causes infections of the skin, lung, bloodstream, and other body parts. Over the past decade,community-acquired methicillin resistant S. aureus (CA-MRSA) infections, which were previously extremely rare, are occurring commonly worldwide. CA-MRSA is the most common cause of skin infection in many locales in the U.S., including Southern California.

CA-MRSA strains are notable for their ability to spread in closed settings and cause recurrent infections among healthy persons. Management of recurrent CA-MRSA infection is challenging and optimal prevention strategies are undefined. Many experts recommend topical agents that decontaminate the body and/or anterior nares. Others suggest environmental decontamination to help control recurrences or transmission within households. However, there are no data that quantify the efficacy and safety of these approaches.

We will conduct a multi-center clinical trial to compare the efficacy and safety of body and environmental decolonization regimens in the prevention of CA-MRSA infection. This trial is being conducted at Kaiser Permanente Southern California (KPSC) sites among KPSC enrollees.

The study population will comprise of persons suffering from recurrent CA-MRSA infection. Household members of this "index subject" will also be offered the chance to enroll in the study. For this clinical trial, all subjects will be randomized in a 2 x 2 design to test: 1) chlorhexidine body washes and nasal mupirocin ointment vs. usual care, and 2) environmental cleansing with ethanol spray and aggressive laundering vs. no environmental cleansing. Household members, should they consent, will also be enrolled into the study into the same treatment arm as "index subjects". We will also perform selected secondary analyses, including studying the efficacy of the interventions at preventing infections in household members. Additionally, we will examine strain relatedness of colonizing and infecting CA-MRSA strains to better understand colonization dynamics within households.

ELIGIBILITY:
Inclusion Criteria:

* Is a member of Kaiser Permanente Southern California (KPSC)
* Have at least 1 culture positive for MRSA in the prior 12 months and at least one skin infection in the prior 12 months. The culture(s) and/or skin infection(s) will:

A. Be associated with mutually exclusive patient encounters that are separated by at least 21 days. The encounters include: outpatient visits to primary care provider; outpatient visits to emergency departments or urgent care facilities; inpatient hospitalizations (admission date is considered the encounter date)

AND

Each patient encounter defined in section A is associated with EITHER:

B. EITHER receipt of a prescription (or course) of antibiotics for a clinical infection.

OR

C. A visit to an outpatient setting (including primary care provider visits, emergency department visits, phone consultations, and urgent care visits) for a skin or skin structure infection.

* Age is 1 month or older
* Ability and willingness to take intranasal medications, topical body washes, and environmental decontamination measures.
* Ability and willingness of subject or legal guardian/representative to give written informed consent.
* Ability and willingness to participate in the study according to treatment allocation even if not randomized to an active intervention.

Exclusion Criteria:

* Current residence in a KPSC-associated chronic care facility or other chronic-care facility (e.g., a rehabilitation facility or nursing home)
* Receipt of hemodialysis or peritoneal dialysis in the prior 12 months
* Any of the following severe underlying conditions: Organ transplantation, active or recent malignancy, cancer, or inflammatory disorder that has required (or would have require treatment) in the prior 12 months, with radiation therapy, surgery, chemotherapy, systemic immunomodulatory therapy (e.g., tumor necrosis factor (TNF)-alpha inhibitors for rheumatic and inflammatory diseases), or corticosteroid therapy (defined as > 7.5 mg prednisone (or equivalent doses of a non-prednisone corticosteroid) daily for adults, or above physiologic levels of prednisone or other corticosteroid therapy daily for children).
* Any of the following major surgical procedure in the prior 12 months: orthopedic procedure, cardiothoracic surgery, or abdominal surgery.
* Use of the following drugs or procedures within 120 days prior to study entry: topical mupirocin (Bactroban or Bactroban Nasal), Chlorhexidine (e.g., Hibiclens or other branded or generic formulations) body washes, or environmental decontamination of the household with ethyl alcohol (e.g., Lysol Brand Disinfectant Spray for Kitchens or other branded or generic formulations), bleach or dilute bleach solutions, or similar regimens
* Current use of systemic antibiotics used specifically to treat skin or skin structure infections, MRSA infections, or S. aureus infections. Patients on systemic therapy noted here must complete the systemic antibiotic therapy prior to enrollment.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Current skin wound or lesion that is deeper than superficial layers of the skin (which is known to be a relative contraindication to topical Hibiclens). Subjects with deeper skin infection may be enrolled when their wound has healed sufficiently so that the wound is no deeper than the superficial skin layers
* Known hypersensitivity or allergic reaction to either topical mupirocin or mupirocin-containing products (e.g., Bactroban or Bactroban Nasal), or chlorhexidine or chlorhexidine-containing (e.g., Hibiclens) topical washes or products containing chlorhexidine.
* Concurrent use of other intranasal products (e.g., saline washes, topical decongestants, antihistamines, or anticholinergics). Patients who use these products who are willing to discontinue therapy for seven days while mupirocin is administered (if they are randomized to this medication) will be allowed to participate in consultation with the patient's provider.
* Chronic skin conditions associated with hypersensitivity to using topical cleansers or preparations.
* Known hypersensitivity among household members to the agents listed above, specifically mupirocin, chlorhexidine, and topical ethanol.
* "Heavy" or excessive use of body decolonizing agents such as triclosan-containing soap or Phisohex, as determined by the Study Site Coordinator.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2007-04; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
A new MRSA or skin infection consistent with MRSA infection. | during the 52-week follow up period

SECONDARY OUTCOMES:
A new skin infection that was cultured and not found to be caused by MRSA. | during the 52-week follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Jared Spotkov, M.D., Principal Investigator — Kaiser Permanente; Loren Miller, M.D., M.P.H., Study Chair — Harbor-UCLA Medical Center (LABiomed)
Locations (6):
- United States (6):
  - Kaiser Permanente, Anaheim, Anaheim, California
  - Kaiser Permanente, Bellflower, Bellflower, California
  - Kaiser Permanente, Harbor City, Harbor City, California
  - Kaiser Permanente, Irvine, Irvine, California
  - Kaiser Permanente, Panorama City, Panorama City, California
  - Kaiser Permanente, West LA, West Los Angeles, California